CLINICAL TRIAL: NCT05539820
Title: The Effect of Distant Reiki on the State Test Anxiety Levels and Exam Success of Nursing Students: A Randomized Controlled Study
Brief Title: Reiki Effects on the State Test Anxiety Levels and Exam Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Medipol University (Other)
Responsible Party: Principal Investigator, NURSEMIN UNAL, Assistant Professor, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 025
Record Dates: First submitted 2022-09-03; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Anxiety; Exam Stress
Keywords: Reiki; Distant Reiki; State Test Anxiety; Exam Success; Nursing Students
MeSH Terms: conditions — Anxiety Disorders | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The students and investigators knew which group they were assigned to. Only the outcome assessor did not know which student was assigned to which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki group (Experimental): PIF-I and STAS were administered to the Reiki group through an online questionnaire. After the pretests of the students were completed, between 14-17 June 2022, the distant reiki application was made under the guidance of a researcher with a Usui Reiki Master &Teacher degree and by the researchers with Reiki -II or Reiki-III degrees. The application was carried out for 20 minutes on four consecutive days. Before the final exams (19 June 2022), the posttests (PIF-II and STAS) were applied to the students through an online questionnaire.
  Interventions: Other: Reiki
- Control Group (No Intervention): PIF-I and STAS were administered to the control group through an online questionnaire. Then before the final exams on 19 June 2022, the posttests (PIF-II and STAS) were applied to the students through an online questionnaire.

INTERVENTIONS:
Other: Reiki — Reiki is based on the belief that disease occurs when an energy center is blocked, and that the energy is transmitted through touch. In distant Reiki, Reiki practitioners followed the traditional Usui Reiki protocol for distant healing. Reiki practitioners first undertake the name of students and then send the healing energy to the students.
  Arms: Reiki group

SUMMARY:
This study aimed to determine the effect of distant Reiki on first-year nursing students' state test anxiety levels and exam success.

DETAILED DESCRIPTION:
Reiki, an energy-based practice based in Japanese culture, consists of the words "rei" meaning "Spirit" and "ki" meaning "universal life force" and means "spiritual directed life force energy". Reiki, accepted as a complementary and alternative therapy (CAM) by the National Center for Complementary and Alternative Medicine, is a simple, natural and safe method that everyone can use; It is a holistic healing method that nourishes the body, mind and spirit. The principle of Reiki is based on the principle that in case of a blockage in an energy center, disease occurs and the energy transferred by touching it strengthens and heals the body's ability to heal itself by opening the blockages. Trained Reiki practitioners can perform the application by holding their hands in certain positions on the recipient's body, as well as remotely. It will also be important for Reiki to become widespread as a nursing practice in many countries, especially for nurse candidates to experience the effects of Reiki on reducing stress and anxiety. In the literature, it is emphasized that uncontrollable test anxiety can also affect the academic success of students. For this reason, it is thought that Reiki, whose effectiveness in coping with stress and anxiety has been demonstrated by various studies, may be effective in coping with exam anxiety of nursing students. A study investigating the effect of Reiki on reducing students' anxiety could not be found in the literature. In this context, it will be the first study to examine the effect of Reiki on reducing anxiety in nursing students.

This randomized controlled prospective study was conducted with first-year nursing students between 10-19 June 2022. The data of the study was collected using "Personal Information Form I-II (PIF)" and "State Test Anxiety Scale (STAS)" via online form. Also, the final exam notes were used for assessing the success of the students, the final exam averages were used.

PIF-I and STAS were applied to the students who met the inclusion criteria and agreed to participate in the study between 10-13 June 2022. Patients were randomized 1:1 into groups by a single therapist according to the block randomization method. There were two arms in the study; Reiki treatment (n=36) and control group (n=35). A second or third-degree Reiki practitioner applied distant Reiki to the students for 20 minutes for four consecutive days (14-17 June 2022) in the Reiki treatment group. In the control group, nothing was done. At 19 June 2022, PIF- II and STAS were applied to all patients.

ELIGIBILITY:
Inclusion Criteria:

* Not having a diagnosed current anxiety disorder or any psychiatric problem,
* Not having a current acute or chronic health problem,
* Willingness to participate in Reiki practice,
* Not having received body-mind therapy (yoga, reiki, meditation, etc.) in the last six months

Exclusion Criteria:

* Those who were diagnosed with an anxiety disorder or a psychiatric illness during the data collection process and need treatment,
* Being Reiki practitioners or trainers,
* Those who refuse to answer the Reiki application and data collection tools,
* Those who want to leave the research while the research is continuing,
* Those who had previously received energy therapies such as Reiki/therapeutic ouch/healing touch and those who used other complementary health practices were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-06-19 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Personal Information Form-I | Baseline.
  There are 16 questions to determine the socio-demographic characteristics of the students (age, gender, marital status, educational status of parents, etc.).
Change from State Test Anxiety Scale | Baseline, 1 day before the exam.
  The scale measured the state test anxiety level of the students. Within the scope of the study, the scale was repeated before the final exams on 19 June 2022. While the minimum score that can be obtained from State Test Anxiety Scale is 22, the maximum score is 88. An increase in the score obtained from the scale means an increase in the level of anxiety.
Personal Information Form-II | 1 day before the exam.
  It was made as a post-test, and it includes 6 questions that question the characteristics of students regarding sleep, tea-coffee-cigarette consumption during the exam period.

CONTACTS AND LOCATIONS:
Overall Officials: Nursemin Ünal, Principal Investigator — Ankara Medipol University
Locations (1):
- Nursemin Ünal, Ankara, None Selected, Turkey (Türkiye)

REFERENCES:
- [Background] Hamaideh SH, Al-Omari H, Al-Modallal H. Nursing students' perceived stress and coping behaviors in clinical training in Saudi Arabia. J Ment Health. 2017 Jun;26(3):197-203. doi: 10.3109/09638237.2016.1139067. Epub 2016 Feb 5. PMID 26850046
- [Background] Bektas Akpinar N, Ozcan Yuce U, Yurtsever S. The Effect of Distant Reiki on the Stress and Fatigue Levels of Nurses Working in COVID-19 Clinics: A Randomized-Controlled, Single-Blind Study. Holist Nurs Pract. 2024 Mar-Apr 01;38(2):102-108. doi: 10.1097/HNP.0000000000000519. Epub 2022 Apr 7. PMID 35435859
- [Background] Chen YW, Hung CH. Predictors of Taiwanese baccalaureate nursing students' physio-psycho-social responses during clinical practicum. Nurse Educ Today. 2014 Jan;34(1):73-7. doi: 10.1016/j.nedt.2013.02.021. Epub 2013 Apr 6. PMID 23566461
- [Background] Torabizadeh C, Bostani S, Yektatalab S. Comparison between the effects of muscle relaxation and support groups on the anxiety of nursing students: A randomized controlled trial. Complement Ther Clin Pract. 2016 Nov;25:106-113. doi: 10.1016/j.ctcp.2016.09.001. Epub 2016 Sep 7. PMID 27863599
- [Background] Cuneo CL, Curtis Cooper MR, Drew CS, Naoum-Heffernan C, Sherman T, Walz K, Weinberg J. The effect of Reiki on work-related stress of the registered nurse. J Holist Nurs. 2011 Mar;29(1):33-43. doi: 10.1177/0898010110377294. Epub 2010 Aug 10. PMID 20699431
- [Background] Diaz-Rodriguez L, Arroyo-Morales M, Fernandez-de-las-Penas C, Garcia-Lafuente F, Garcia-Royo C, Tomas-Rojas I. Immediate effects of reiki on heart rate variability, cortisol levels, and body temperature in health care professionals with burnout. Biol Res Nurs. 2011 Oct;13(4):376-82. doi: 10.1177/1099800410389166. Epub 2011 Aug 5. PMID 21821642
- [Background] Asturias N, Andrew S, Boardman G, Kerr D. The influence of socio-demographic factors on stress and coping strategies among undergraduate nursing students. Nurse Educ Today. 2021 Apr;99:104780. doi: 10.1016/j.nedt.2021.104780. Epub 2021 Jan 20. PMID 33516979